CLINICAL TRIAL: NCT07394517
Title: Efficacy of Phospholipid Omega-3 (Ruby-O) Versus Conventional Omega-3 on the Omega-3 Index in Patients With Mixed Dyslipidemia: A 24-Week Randomized, Double-Blind, Parallel Trial
Brief Title: ATLANTIS Trial: Phospholipid Omega-3 Versus Conventional Omega-3
Acronym: ATLANTIS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación del Caribe para la Investigación Biomédica (Other)
Collaborators: Naturmega (Unknown)
Responsible Party: Principal Investigator, Miguel Urina-Triana PhD, Principal Investigator, Fundación del Caribe para la Investigación Biomédica
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIOS-ATLANTIS-01
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Mixed Dyslipidemia
Keywords: Mixed dyslipidemia; Omega -3 Index; Phospholid omega-3; Triglycerides; EPA; DHA; Dietary Suplement; Cardiovascular Risk

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, parallel-group study with three arms comparing two dose levels of a phospholipid omega-3 supplement versus a conventional triglyceride omega-3 formulation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All study products are identical in appearance, packaging, and labeling to maintain masking of participants, investigators, care providers, and outcome assessors throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ruby-O Moderate Dose (Experimental): Participants receive a phospholipid-based omega-3 supplement (Ruby-O) providing approximately 995 mg of EPA+DHA daily, administered orally once daily with meals for 24 weeks.
  Interventions: Dietary Supplement: Phospholipid Omega-3
- Ruby-O High Dose (Experimental): Participants receive a phospholipid-based omega-3 supplement (Ruby-O) providing approximately 1491 mg of EPA+DHA daily, administered orally once daily with meals for 24 weeks.
  Interventions: Dietary Supplement: Phospholipid Omega-3
- Conventional Omega-3 (Experimental): Participants receive a conventional triglyceride-based omega-3 supplement providing EPA 900 mg and DHA 600 mg daily, administered orally once daily with meals for 24 weeks.
  Interventions: Dietary Supplement: Triglyceride Omega-3

INTERVENTIONS:
Dietary Supplement: Phospholipid Omega-3 — Phospholipid-based omega-3 dietary supplement containing eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), administered orally once daily with meals for 24 weeks at a moderate dose level.
  Arms: Ruby-O High Dose
Dietary Supplement: Phospholipid Omega-3 — Phospholipid-based omega-3 dietary supplement containing eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), administered orally once daily with meals for 24 weeks at a higher dose level.
  Arms: Ruby-O Moderate Dose
Dietary Supplement: Triglyceride Omega-3 — Conventional triglyceride-based omega-3 dietary supplement containing eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), administered orally once daily with meals for 24 weeks.
  Arms: Conventional Omega-3

SUMMARY:
This study is a clinical trial designed to compare two forms of omega-3 supplements in adults with mixed dyslipidemia. Mixed dyslipidemia is a condition in which blood fat levels, such as triglycerides and cholesterol, are not within the recommended range and may increase the risk of cardiovascular disease.

Participants in this study will be randomly assigned to receive one of three study products: a phospholipid-based omega-3 supplement (Ruby-O) at a moderate dose, the same phospholipid-based omega-3 supplement at a higher dose, or a conventional omega-3 supplement in triglyceride form. All study products will be taken by mouth once daily with food for 24 weeks.

The main goal of the study is to evaluate changes in the Omega-3 Index, a blood test that reflects the amount of omega-3 fatty acids incorporated into red blood cell membranes. Additional goals include evaluating changes in blood lipid levels, markers of inflammation, blood sugar metabolism, body weight, blood pressure, treatment adherence, and safety.

This study is sponsored by the Fundación del Caribe para la Investigación Biomédica and is conducted in adults who are receiving stable statin therapy. Participation in the study is voluntary, and all participants may withdraw at any time.

DETAILED DESCRIPTION:
Mixed dyslipidemia is a metabolic condition characterized by elevated triglyceride levels and other lipid abnormalities and is associated with increased residual cardiovascular risk despite standard lipid-lowering therapy. Addressing lipid abnormalities beyond low-density lipoprotein cholesterol may help reduce this residual risk.

The Omega-3 Index is defined as the percentage of eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) in erythrocyte membranes and reflects long-term omega-3 fatty acid exposure and tissue incorporation. Higher Omega-3 Index values have been associated with more favorable cardiovascular risk profiles.

The chemical form of omega-3 fatty acids influences their absorption and bioavailability. Phospholipid-bound omega-3 formulations have demonstrated more efficient intestinal absorption and cellular membrane incorporation compared with conventional triglyceride-based formulations. This study was designed to evaluate whether different dose levels of a phospholipid-based omega-3 supplement result in greater changes in the Omega-3 Index compared with a conventional triglyceride-based omega-3 supplement.

This is a randomized, double-blind, parallel-group clinical trial with three study arms. Eligible participants are adults with mixed dyslipidemia receiving stable statin therapy. Participants are randomly assigned to receive either a phospholipid-based omega-3 supplement at a moderate dose, the same supplement at a higher dose, or a conventional omega-3 supplement in triglyceride form. All study products are administered orally once daily with food for a total duration of 24 weeks.

The primary objective of the study is to compare the Omega-3 Index at week 24 among treatment groups, adjusted for baseline values. Secondary objectives include evaluation of changes in lipid parameters, inflammatory biomarkers, glucose metabolism, anthropometric measures, blood pressure, treatment adherence, and safety outcomes.

The study is conducted in accordance with ethical principles for research involving human participants and has been approved by an institutional ethics committee. Participation is voluntary, and all participants provide written informed consent prior to any study-related procedures.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:
* Adults aged 18 years or older.
* Diagnosis of mixed dyslipidemia.
* Fasting triglyceride levels between 135 and 499 mg/dL.
* Body mass index (BMI) ≥27 kg/m².
* High-sensitivity C-reactive protein (hs-CRP) >2 mg/L.
* Stable statin therapy for at least 8 weeks prior to enrollment.
* Ability and willingness to provide written informed consent.

Exclusion Criteria:

* Fasting triglyceride levels ≥500 mg/dL.
* History of a recent cardiovascular event.
* Significant hepatic or renal disease.
* Pregnancy or breastfeeding.
* Known allergy or hypersensitivity to fish or seafood.
* Use of omega-3 supplements within 8 weeks prior to randomization.
* Participation in another interventional clinical trial within 8 weeks prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Omega-3 Index (O3I) | Week 24
  The Omega-3 Index (O3I) is a continuous biochemical measure defined as the percentage of eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) in erythrocyte membranes, measured by standardized erythrocyte fatty acid analysis. It is expressed as a percentage (%), with values observed in adult populations typically ranging from approximately 2% (very low levels) to 15% (very high levels), although no absolute theoretical maximum is defined. Higher Omega-3 Index values indicate a more favorable cardiovascular risk profile. The primary analysis uses the value at week 24, adjusted for baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundación del Caribe para la Investigación Biomédica (Fundación BIOS), Barranquilla, Atlántico, Colombia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study does not include a formal data-sharing plan and to protect participant privacy and confidentiality, in accordance with the informed consent and applicable data protection regulations.

REFERENCES:
- [Background] Harris WS, Von Schacky C. The Omega-3 Index: a new risk factor for death from coronary heart disease? Prev Med. 2004 Jul;39(1):212-20. doi: 10.1016/j.ypmed.2004.02.030. PMID 15208005